CLINICAL TRIAL: NCT04563650
Title: Kinetics of COVID-19-neutralising Antibodies in Patients Residing in EHPAD / USLD: Influence of Immunosenescence
Brief Title: COVID-19 Serology and Immunosenescence
Acronym: SERO-CoV-OLD
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: PI2020_843_0079
Record Dates: First submitted 2020-09-18; First posted 2020-09-24 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Covid19; Geriatric Medicine; Seroconversion; Immunosenescence
Keywords: Covid19; geriatric medicine; seroconversion; immunosenescence
MeSH Terms: conditions — COVID-19; HIV Seropositivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID-19 positive resident (Experimental)
  Interventions: Biological: blood sample
- COVID-19 negative resident (Active Comparator)
  Interventions: Biological: blood sample

INTERVENTIONS:
Biological: blood sample — Sample collection of 4 to 10 tubes of whole blood will be done according to centre Saint-Victor's protocol.

SUMMARY:
This study aims to determine how long COVID-19 neutralizing antibodies can be detected in an elderly institutionalized population presenting fragility factors.

This study also aims to stratify seroconversion by immunological profiles of the elderly patients residing in the EHPAD. This stratification requires the measurement of immunological marker levels already described in immunosenescence and also involved in the development of certain chronic infectious diseases more common in the elderly population. This analysis will enable the investigators to describe an immunological, clinical and biological profile representing a patient who has developed an immunity against COVID 19. It will also help the investigators to understand the different mechanisms leading to a reduced immune response after a potential administration of a vaccine. Finally, it will help describe the immune profiles of elderly residents who presented with non-severe forms of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Residents of the EHPAD/USLD St Victor of the Amiens CHU who took part in the screening campaign (RT-PCR and serology) organized by the Amiens CHU
* residents who signed a consent form to participate in the study

Exclusion Criteria:

* The patient or his legal representative refused to participate in the study
* Heavily sedated patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2020-09-18 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
titers of COVID-19 neutralising antibodies | day 0
titers of COVID-19 neutralising antibodies | at 3 months
titers of COVID-19 neutralising antibodies | at 6 months
titers of COVID-19 neutralising antibodies | at 9 months

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No